CLINICAL TRIAL: NCT03639974
Title: Expiratory Positive Pressure With Blow-bottle Device Versus Expiratory Positive Airway Pressure (EPAP) in Patients After Postoperative Cardiac Surgery: Randomized Clinical Trial
Brief Title: Positive Expiratory Pressure With Blow-bottle Device Versus EPAP After Postoperative Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: UNIVERSIDADE FEDERAL DO RIO GRANDE DO SUL (UFRGS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0460
Record Dates: First submitted 2018-07-13; First posted 2018-08-21 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial that will be performed according to the CONSORT Statement (Consolidated Standards of ReportingTrials).
Who Masked: Outcomes Assessor
Masking Description: Double blind: allocation concealment and outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PEP in a blow-bottle device (Active Comparator): Blow-bottle device of 10cmH2O.
  Interventions: Other: PEP in a blow-bottle device
- EPAP Positive airway expiratory pressure (Active Comparator): EPAP with pressure of 10 cmH2O.
  Interventions: Other: EPAP
- conventional physiotherapy (Sham Comparator): Ventilatory exercises, bronchial hygiene techniques, exercises for upper and lower limbs (previous motor condition) stretching, orientation and walking.
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: PEP in a blow-bottle device — A 500-milliliter enteral nutrition vial will be used, which will contain a hole in the side, where two silicone tubes of 20 centimeters long will be inserted together with tape on the bottleneck of the vial. To perform the exercise, the vial will be filled with water leaving a water column of 10 cm high. Deep inspirations will be requested at a volume greater than the tidal volume and less than the total lung capacity that can be performed via nasal or oral, then with the mouth connected to the extensors, the patient will exhale slowly, avoiding to totally empty the lungs. The protocol will be executed twice a day, three sets of ten repetitions. The group will receive the conventional physiotherapy of the cardiac intensive care unit of the HCPA.
  Arms: PEP in a blow-bottle device
Other: EPAP — The Vital Signs ® EPAP kit will be used. Exercises will be performed in the bed, and as soon as the patient is released by the medical team to leave the bed, they can be performed in the sitting position or in orthostasis. For performing the exercise, the EPAP mask will be connected to the face of the patient. The expiratory pressure will be adjusted to 10cmH2O. Deep inspirations will be requested at a volume greater than the tidal volume and below the total lung capacity, then the patient will exhale slowly. The protocol will be executed twice a day, three sets of ten repetitions. The group will receive the conventional physiotherapy of the cardiac intensive care unit of the HCPA, as described in the conventional physiotherapy group.
  Arms: EPAP Positive airway expiratory pressure
Other: conventional physiotherapy — Conventional physical therapy consists of ventilatory exercises, bronchial hygiene techniques, passive, active-assisted or active exercises for upper and lower limbs, and resisted lower limb exercises; stretching, cough and walking guidelines. Initially the exercises will be performed in the bed, as soon as this is withdrawn and the patient is released by the medical team to leave the bed, the progression of the exercises to be performed in the sitting position, orthostasis, and ambulation is performed, this usually occurs on the 2nd postoperative day, after the removal of the mediastinal drain . Under supervision of the physiotherapist, the protocol will be performed twice daily, two sets of ten repetitions.
  Arms: conventional physiotherapy

SUMMARY:
Cardiac surgery is a recommended therapeutic option as a form of secondary prevention for the treatment of cardiovascular diseases, but may present postoperative alterations such as reduction of pulmonary volumes and flows, impairment in gas exchange and increase in the rate of pulmonary complications. The use of positive pressure may reduce these complications. Objective: To evaluate the efficacy of positive expiratory pressure (PEP) in the blow-bottle device compared to expiratory positive airway pressure (EPAP), both associated with conventional physiotherapy, and conventional physiotherapy in the pulmonary function in postoperative cardiac patients through a randomized clinical trial. Methods: The study was approved by the Research Ethics Committee of the Hospital de Clínicas of Porto Alegre (CAEE: 70213617.6.0000.5327). Patients undergoing cardiac surgery were randomized into three groups: positive expiratory pressure with blow-bottle device associated with conventional physiotherapy (G1), positive expiratory pressure in the airways with unidirectional valve associated with conventional physiotherapy (G2), and the third group only the conventional physiotherapy of HCPA cardiac intensive care unit (G3). Initially, an evaluation was performed through spirometry, manovacuometry, radiological changes in the preoperative period, prior to the interventions (immediate postoperative) and on the third postoperative day, immediately prior to cardiac intensive care unit discharge. Pulmonary complications were assessed on the third postoperative day, and length of stay (at the Intensive Care Unit and hospital) were recorded untill discharge.

DETAILED DESCRIPTION:
Cardiac surgery is a recommended therapeutic option as a form of secondary prevention for the treatment of cardiovascular diseases, but may present postoperative alterations such as reduction of pulmonary volumes and flows, impairment in gas exchange and increase in the rate of pulmonary complications. The use of positive pressure may reduce these complications. Objective: To evaluate the efficacy of positive expiratory pressure (PEP) in the blow-bottle device compared to expiratory positive airway pressure (EPAP), both associated with conventional physiotherapy, and conventional physiotherapy in the pulmonary function in postoperative cardiac patients. Methods:This is a randomized clinical trial, with patients in postoperative cardiac surgery. On the first day of postoperative, the patients will be randomized into three groups: 1 group that will receive positive expiratory pressure with blow-bottle device associated with conventional physiotherapy; 2- group that will receive positive expiratory pressure in the airways with valve unidirectional therapy associated with conventional physiotherapy; 3- group that will only receive conventional physiotherapy. The intervention of the positive expiratory pressure with blow-bottle device group will consist of exercise with a blow-bottle device of 10 cm high; the positive expiratory pressure in the airways group, exercise with unidirectional positive expiratory pressure valve (10cmH2O). Both the groups will perform three sets of 10 repetitions per day, by the third day of PO. The third group will receive conventional physiotherapy of intensive care unit. The outcomes evaluated will be: pulmonary function (primary), respiratory muscle strength, pulmonary complications, radiological changes and length of stay (at the Intensive CareUnit - ICU - and hospital). Assessment of pulmonary function, muscle strength and radiological changes will be performed in the preoperative period, prior to the interventions and on the third postoperative day, immediately prior to discharge of cardiac intensive care unit. Pulmonary complications and ICU length of stay will be recorded after discharge from intensive care unit cardiac. The length of hospital stay was recorded after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

Elective cardiovascular surgery of:

coronary artery bypass graft surgery alone

coronary artery bypass graft surgery combined with aortic valve surgery

coronary artery bypass graft surgery combined with bicuspid valve surgery

coronary artery bypass graft surgery combined with tricuspid valve surgery

Aortic valve surgery

Bicuspid valve surgery

Tricuspid valve surgery

All on spontaneous ventilation or with supplemental oxygen support.

Exclusion Criteria:

Patients with hemodynamic instability (heart rate> 120bpm, clinically important hypotension - vasopressor dose ≥ 0.1mcg / kg / min)

Cardiac arrhythmia

Heart transplantation

Angina at rest and/or minor efforts

Mechanical ventilation for more than 24 hours

Re-hospitalized patients with decompensated heart failure

Noninvasive mechanical ventilation

Non-collaborative and with cognitive inability to understand the procedures

Reintubated patients

Re-operated patients

In order to perform the pulmonary function test, patients may not present the following contraindications:

hemoptysis

recent angina

retinal detachment

hypertensive crisis

pulmonary edema

thoracic aortic aneurysm

In order to perform the respiratory muscle strength test, patients may not present the following contraindications:

acute myocardial infarction

recent unstable angina

severe and uncontrolled systemic arterial hypertension

aortic aneurysm

pneumothorax

pleurocutaneous or pulmonary fistulas

surgery or recent trauma to the upper airways, chest or abdomen

abdominal hernia

acute middle ear problems

glaucoma or retinal detachment

hydrocephalus

meningocele

neurological processes that favor the choking of tonsils

general state of physical or mental impairment that impedes the patient's collaboration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Pulmonary function - forced vital capacity | three days
  Pulmonary function through spirometry. Spirometry allows to measure forced vital capacity. It's the air volume expired, quickly, after an inspiration deep maximum.
Pulmonary function - forced expiratory volume in the first second | three days
  Pulmonary function through spirometry, that allows to measure forced expiratory volume in the first second. It's the maximum expired volume at the first second of an maximum expiration .
Pulmonary function - the ratio: forced expiratory volume in the first second / forced vital capacity | three days
  Pulmonary function through spirometry, obtained through forced maneuver (forced vital capacity) and forced expiratory volume in the first second - represents the maximum expired volume at the first second of an maximum expiration.

SECONDARY OUTCOMES:
Respiratory muscle strength - maximum expiratory pressure | three days
  Performed through a manometer in step cmH2O, of the brand Globalmed model MV300. Maximum expiratory pressure.
Respiratory muscle strength - maximal inspiratory pressure | three days
  Performed through a manometer in step cmH2O, of the brand Globalmed model MV300. Maximal inspiratory pressure will be measured.
Pulmonary complications - atelectasis | three days
  According to the definitions of the European Journal of Anaesthesiology
Pulmonary complications - pleural effusion | three days
  According to the definitions of the European Journal of Anaesthesiology
Pulmonary complications - pneumothorax | three days
  According to the definitions of the European Journal of Anaesthesiology
Pulmonary complications - pneumonia | three days
  According to the definitions of the European Journal of Anaesthesiology
Pulmonary complications - respiratory infection | three days
  According to the definitions of the European Journal of Anaesthesiology
Pulmonary complications - respiratory failure | three days
  According to the definitions of the European Journal of Anaesthesiology
Radiological changes - pleural effusion | three days
  rated on chest X-ray, according to the scale proposed by Staton et al.
Radiological changes - atelectasis | three days
  rated on chest X-ray, according to the scale proposed by Staton et al.
Radiological changes - consolidation | three days
  rated on chest X-ray, according to the scale proposed by Staton et al.
Radiological changes - pneumothorax | three days
  rated on chest X-ray, according to the scale proposed by Staton et al.
Radiological changes - pulmonary edema | three days
  rated on chest X-ray, according to the scale proposed by Staton et al.
Length of Intensive Care Unit (ICU) stay | three days
  Length of ICU stay (days) search electronic records
Length of hospital stay | up to 25 days
  Length of hospital stay (days) search electronic records

CONTACTS AND LOCATIONS:
Overall Officials: Graciele Sbruzzi, doctor, Principal Investigator — HCPA
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pieczkoski SM, de Oliveira AL, Haeffner MP, Azambuja ACM, Sbruzzi G. Positive expiratory pressure in postoperative cardiac patients in intensive care: A randomized controlled trial. Clin Rehabil. 2021 May;35(5):681-691. doi: 10.1177/0269215520972701. Epub 2020 Nov 24. PMID 33233946